CLINICAL TRIAL: NCT01570452
Title: Matrilysin Expression in Different Stages of Colorectal Tumors
Acronym: MMP7
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Polistena MD, MD specialist in General Surgery, University of Roma La Sapienza
Other Study IDs: andreapolistena1
Record Dates: First submitted 2012-03-31; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Colorectal Cancer Stage 0; Colorectal Cancer Stage I; Colorectal Cancer Stage II; Colorectal Cancer Stage III; Colorectal Cancer Stage IV
Keywords: matrilysin; MMP-7; colorectal cancer; adenoma; lymph nodes
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — normal mucosa, cancer tissue, lymph nodes and serum from cancer patients serum from healty volunteers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- healthy volunteers: healthy subjects not affected by benign or malignant colonic disease
  Interventions: Procedure: colonic or colorectal resection
- benign colonic tumor patients: patients affected by benign colonic tumor such as adenoma
  Interventions: Procedure: colonic or colorectal resection
- cancer patient I-II stage: Patients affected by colonic cancer in I-II stage
  Interventions: Procedure: colonic or colorectal resection
- cancer patients III-IV stage: Patients affected by colonic cancer in III-IV stage
  Interventions: Procedure: colonic or colorectal resection

INTERVENTIONS:
Procedure: colonic or colorectal resection — standard laparotomic resection of colon-rectum including right hemicolectomy, left hemicolectomy, sigmoidectomy, anterior resection

SUMMARY:
Matrix metalloproteinases (MMPs) have been shown to be involved in cancer biology. Significant expression of MMP-7 (matrilysin) in colorectal cancer is mainly associated with metastatic disease even though it is expressed in most tumor states. Our purpose is to analyse MMP-7 in bowel and lymph nodes of different tumor stages and to evaluate its expression as a potential biomarker of cancer disease in patients surgically treated for benign and malignant colorectal tumors. Tumoral tissue, lymph nodes and serum samples from recruited Patients plus serum samples from healthy volunteers are analysed for matrilysin expression by histology, immunohistochemistry, ELISA and Western blotting.

If Matrilysin increases with increasing dysplasia and cancer disease stage in tumor tissue as well as in the regional lymph nodes it might be used as a complement in investigating suspected locally advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* benign colonic neoplasm not suitable for endoscopic treatment,
* malignant colonic neoplasm with indication to primary surgical treatment

Exclusion Criteria:

* neo-adjuvant radiotherapy,
* chemo-radiotherapy,
* language problems and withdrawal of consent

Ages: 40 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients affected by colorectal neoplasm admitted to our department of surgery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Polistena, MD, Principal Investigator — Department of Surgery Pietro Valdoni, University La Sapienza Rome
Locations (1):
- Departement of Surgery Pietro Valdoni, Rome, Italy

REFERENCES:
- [Background] Mori M, Barnard GF, Mimori K, Ueo H, Akiyoshi T, Sugimachi K. Overexpression of matrix metalloproteinase-7 mRNA in human colon carcinomas. Cancer. 1995 Mar 15;75(6 Suppl):1516-9. doi: 10.1002/1097-0142(19950315)75:6+3.0.co;2-7. PMID 7889484